CLINICAL TRIAL: NCT04739553
Title: His Pacing in Patients Without Need for Cardiac Resynchronization - Clinical Feasibility and Cardiac Electrical Activation
Brief Title: His Pacing Feasibility and Cardiac Electrical Activation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Anna Margrethe Thoegersen, Medical Doctor, Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-20200032
Record Dates: First submitted 2021-01-19; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Pacing-Induced Cardiomyopathy; AV Block; Heart Failure
MeSH Terms: conditions — Atrioventricular Block; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- His Pacing (Experimental): Implant of a supplementary His pacing lead in addition to a traditional RV pacing lead.
  Interventions: Device: His Pacing

INTERVENTIONS:
Device: His Pacing — The patients will receive a pacemaker implant with a traditional right ventricular pacing lead and an additional His pacing lead in a basal high septal position at the level of the proximal electrical conduction system (His). An atrial lead is implanted if dual chamber pacing is needed. All leads are connected to a biventricular pacemaker with the His lead in the LV port.

SUMMARY:
This study will examine the clinical feasibility of His pacing in patients with expected high demand for ventricular pacing and no established indication for cardiac resynchronization therapy. Secondarily, examine differences in electrical and mechanical cardiac activation between traditional pacing and His pacing.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all eligible patients giving written consent will be included. The study is a clinical single-center interventional study. The patients (n = 25) need to have an expected high demand for ventricular pacing and no established class I indication for cardiac resynchronization therapy. They will receive a pacemaker implant with a traditional right ventricular pacing lead and an additional His pacing lead in a basal high septal position at the level of the proximal electrical conduction system (His). An atrial lead is implanted if dual chamber pacing is needed. All leads are connected to a biventricular pacemaker with the His lead in the LV port. Postoperatively, the baseline examinations will include: transthoracic echocardiography, 12-lead ECG with a 3D photography of the chest wall to document ECG electrode location, and a contrast-enhanced cardiac CT scan. The echocardiography and ECG will be performed during traditional right ventricular pacing only and His pacing only. His pacing will be used as the permanent programming of choice if feasible during follow up. The CT scan is used for documenting the final positions of the pacing leads and to create a patient-specific 3D model of the cardiac electrical activation using a software which enables merging of a CT scan and ECG and a CT chest photography. During follow up (1-3 and 12 months), transthoracic echocardiography, 12-lead ECG and 3D chest photography are repeated for assessment of mechanical and electrical function during pacing. The performance of all implanted pacing lead will be evaluated at each follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Permanent pacemaker indication with expected high demand of right ventricular pacing (>40%) and left ventricular ejection fraction >40%.

Exclusion Criteria:

* No class I indication for CRT pacemaker (HRS 2018 Pacing Guidelines)
* Hemodynamically unstable patients
* Severely reduced kidney function
* Former serious adverse reactions to contrast media
* Pregnant or lactating
* Severe psychiatric disorder which can compromise compliance with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Rate of chronic His pacing success | Evaluated at 1 year follow up
  Chronic His capture with clinically acceptable pacing threshold (<=3.5V)

SECONDARY OUTCOMES:
Rate of perioperative His pacing success | The implant procedure duration i.e. incision to skin closure
  Perioperative his capture with clinically acceptable pacing threshold (<=3.5V)
QRS duration (ms) | Implantation to 1 year follow up
  Comparing His pacing and RV pacing
Changes in left ventricular echocardiographic two-dimensional strain dyssynchrony parameters | Implant to 1 year follow up
  Comparing left ventricular mechanical dyssynchrony during His pacing and RV pacing using echocardiographic two-dimensional longitudinal strain
Changes in regional right and left ventricular electrical activation delay | Implant to 1 year follow up
  Comparing electrical activation pattern during His pacing and RV pacing using non-invasive electroanatomical mapping. This is achieved using software that merges data from a 12-lead electrocardiogram (ECG), chest wall three-dimensional picture of ECG lead positions, and a cardiac computed tomography scan.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Riahi, MD PhD, Study Director — Aalborg University Hospital; Peter Søgaard, MD DMSc, Study Director — Aalborg University Hospital

IPD SHARING:
Plan to Share IPD: No